CLINICAL TRIAL: NCT01966484
Title: Low Dose Mivacurium vs. Low Dose Succinylcholine for Rigid Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSK003
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Intubating Conditions; Performance With Respiratory Exercise Device; Postoperative Myalgia
Keywords: Succinylcholine; Mivacurium; Rigid Bronchoscopy; Intubating conditions; Short Procedure
MeSH Terms: interventions — Succinylcholine; Mivacurium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Succinylcholine (Active Comparator): Patient receive succinylcholine as a muscle relaxant (0,5mg/kg) after induction of general anaesthesia for rigid bronchoscopy.
  Interventions: Drug: Succinylcholine
- Mivacurium (Active Comparator): Patients receive mivacurium (0,08mg/kg) as a muscle relaxant after induction of general anaesthesia for rigid bronchoscopy. At the end of the procedure and a twitch of 25% mivacurium was reversed with neostigmine (50 microg/kg) and atropin (10 microg/kg)
  Interventions: Drug: Mivacurium

INTERVENTIONS:
Drug: Succinylcholine — Anaesthesia was induced and maintained with propofol(1-2mg/kg and 5mg/kg/h) and remifentanil (1µg/kg and 0,2µ/kg/min). The study arm is immobilized and a dual electrode for peripheral nerve stimulation is placed over the ulnar nerve near the wrist. Neuromuscular monitoring is performed with accelerometry. the patients receive the muscle relaxant according to the study group.
  Other Names: Mivacurium; Rigid Bronchoscopy
  Arms: Succinylcholine
Drug: Mivacurium — Anaesthesia was induced and maintained with propofol(1-2mg/kg and 5mg/kg/h) and remifentanil (1µg/kg and 0,2µ/kg/min). The study arm is immobilized and a dual electrode for peripheral nerve stimulation is placed over the ulnar nerve near the wrist. Neuromuscular monitoring is performed with accelerometry. the patients receive the muscle relaxant according to the study group.
  Other Names: Succinylcholine; Rigid Bronchoscopy
  Arms: Mivacurium

SUMMARY:
Succinylcholine is commonly used for neuromuscular relaxation for short procedures such as rigid bronchoscopy. A alternative is the application of low dose mivacurium, reversed with neostigmine. The investigators compare the intubating conditions, incidence of postoperative myalgia (POM), patient satisfaction and the postoperative performance with respiration exercise device for these two muscle relaxants.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yr
* scheduled for elective rigid bronchoscopy

Exclusion Criteria:

* known neuromuscular disease
* significant hepatic or renal dysfunction
* family history of malignant hyperthermia
* known allergy to one of the drugs used in this protocol
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Intubating condition | After induction of general anaesthesia (after 3-5 minutes)
  For measuring the intubation conditions the scoring system proposed for Good clinical Research Practice using the following variables is used: conditions of inserting the rigid bronchoscope, vocal cord position and coughing

SECONDARY OUTCOMES:
Postoperative Myalgia | 72 hours after intervention
  The severity of POM was measured using a four point scale:
  0=no myalgia
  1. minor pain limited to one area of the body
  2. muscle pain or stiffness noticed spontaneously by the patient, which may have required analgesic therapy
  3. generalized, severe or incapacitating discomfort
postintervention performance with a expiration exercise device | 72 hours after intervention
  The performance with a respiration exercise device, which measures the expirational volume, before and after intervention.

OTHER OUTCOMES:
Patient satisfaction | 72 hours after intervention
  Measurement on a numeric ten point scale (10=totally satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Grietje Beck, Prof, Study Chair — Dr. Horst Schmidt Klinik GmbH 65199 Wiesbaden, Germany
Locations (1):
- Dr. Horst Schmidt Klinik GmbH, Wiesbaden, Germany